CLINICAL TRIAL: NCT05038215
Title: Increasing Adherence to Oral Appliance Therapy for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020H0406
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea; Adherence, Patient
Keywords: multifactor intervention; oral appliances
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Intervention Model Description: To determine if the interventions increase adherence in the experimental group compared with a control group receiving the standard protocol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After recruitment and informed consent are complete, subjects will be randomized to the control or experimental group using Random.org. This is a true random number service that generates randomness via atmospheric noise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multifactor intervention (Experimental): The experimental group will receive adherence promotion techniques in addition to routine care.
  Interventions: Behavioral: adherence promotion techniques
- Control (Active Comparator): The control group will receive routine care
  Interventions: Procedure: Routine Care

INTERVENTIONS:
Behavioral: adherence promotion techniques — The experimental group will receive adherence promotion techniques in addition to routine care, including 1-additional information tailored for the spouse/partner, persons living with the patient. 2- Educational material delivered at follow up appointments and by mail at intervals agreed upon by the patient and the clinician. 3- Electronic reminder/communication system established by patient and provider. 4-Follow up communication from the dental provider of the oral appliance to the primary care physician and with patient's approval, their general dentist. 5- After the 3 month follow up visits the patient will be provided with reports about their appliance wear per week. 6-Gift card delivery, $25, at 6 month follow up if a follow up with sleep physician is scheduled.
  Arms: multifactor intervention
Procedure: Routine Care — The control group will receive routine care
  Arms: Control

SUMMARY:
Obstructive sleep apnea is a chronic condition that has serious health consequences including increased risk of hypertension, type-2 diabetes, heart disease, stroke and reduced life expectancy. This study proposes to use behavioral reinforcement and support to increase adherence to oral appliance therapy for obstructive sleep apnea. The control group in the study will receive routine care. In addition, their oral appliance wear time will be monitored using a sensor built into the appliance. Routine care includes an initial 1-hr consult, then delivery of the oral appliance (with sensor) and follow-up appointments at 1 week, 1 month, 3 months, 6 months, and 1 year. The second, experimental group will receive adherence promotion techniques in addition to routine care. These adherence promotion techniques can be categorized into 6 methods. 1- spouse/partner included in a patient counseling session. 2- Educational brochure delivery at follow up appointments. 3- Electronic reminder/communication system established by patient and provider. 4-Follow up communication between primary care physician and orthodontist. 5-Celebratory certificate for good adherence with the oral appliance evaluated at 3 month, and 6 month visits. 6-Gift card delivery, $25, when patient schedules a follow up with sleep physician. Patients will be followed for within the research protocol for 6 months. There are no additional risks involved with the research and the anticipated benefit is to develop methods to increase adherence to treatment for obstructive sleep apnea. This will benefit many patients with obstructive sleep apnea who use oral appliances to control the condition.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants must have a diagnosis of OSA and have been referred for an oral appliance to treat this condition. The participants must have no past experience with oral appliances. Patients must be able to read and converse in English.

Exclusion Criteria:

* Participants who cannot read English will be excluded because all educational material in the study is in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
A multifactorial intervention in addition to standard care increases adherence rates in patients using a titratable oral appliance to treat obstructive sleep apnea (OSA) | 6 months
  The experimental interventions resulted in statistically significant improvements in patient adherence to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Faculty Practice, Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No